CLINICAL TRIAL: NCT00868166
Title: Phase II/III, Multicenter, Randomized, Parallel Group, Double-blind, Placebo Controlled Study to Assess Safety and Efficacy of TRO19622 in Amyotrophic Lateral Sclerosis (ALS) Patients Treated With Riluzole
Brief Title: Safety and Efficacy of TRO19622 as add-on Therapy to Riluzole Versus Placebo in Treatment of Patients Suffering From ALS
Acronym: MITOTARGET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: WN29853; EudraCT Number:2008-007320-25; TRO19622 CL E Q 1015-1 (Other: trophos id)
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; TRO19622; Trophos
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — olesoxime; Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olesoxime (Experimental): 2 Capsules of TRO19622 (330mg) once a day with the noon meal as add-on therapy to riluzole 50mg bid
  Interventions: Drug: Olesoxime; Drug: Riluzole
- Placebo Comparator (Placebo Comparator): 2 Capsules of Placebo once a day with the noon meal as add-on therapy to riluzole 50mg bid
  Interventions: Drug: Placebo Comparator; Drug: Riluzole

INTERVENTIONS:
Drug: Olesoxime — 2 capsules of TRO19622 (330mg) once a day with the noon meal as add-on therapy to riluzol 50mg bid
  Other Names: TRO19622
  Arms: Olesoxime
Drug: Placebo Comparator — 2 capsules of Placebo once a day with the noon meal as add-on therapy to riluzole 50mg bid
  Other Names: Placebo
  Arms: Placebo Comparator
Drug: Riluzole — Riluzole given as add-on therapy 50mg bid
  Other Names: Rilutek

SUMMARY:
The purpose of the assay is to assess the safety and the efficacy of TRO19622 330 mg QD as add-on therapy to riluzole 50 mg bid in the treatment of patients suffering from ALS, as compared to placebo, assessed by the 18-month survival rate.

DETAILED DESCRIPTION:
A stand alone treatment with TRO19622 is not acceptable for ethical reasons. Riluzole is an approved and widely used ALS treatment in the European community, in Japan and in the USA.

Therefore, in this study, TRO19622 will be assessed as add-on to riluzole in patients suffering from ALS.

At the start of the study, patients will be randomized to one of two groups : TRO19622 (330 mg QD or placebo (once a day).

Each treatment will be administered for 18 months under double-blind conditions. The product under evaluation will be administered to patients receiving the standard of care for ALS, including riluzole.

Riluzole dosage (50 mg bid) must be stable and well tolerated for at least one month prior to inclusion into the study.

After the double-blind period, open-label administration of TRO19622 will be allowed for safety and survival assessments and until efficacy results are available.

A separate open-label protocol will be written 6 months after the randomization of the last patient into the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sporadic or familial Amyotrophic Lateral Sclerosis
* Patients with a clinical diagnosis of laboratory-supported probable, probable, or definite ALS according to the modified El Escorial criteria8.
* Have signed an Informed Consent to participate to the trial before any study related procedure has taken place.
* Be of age >18 (exclusive) and < 80 years (inclusive).
* If a female, not lactating, has a negative pregnancy test and agrees to use an effective method of birth control.
* Onset of ALS Symptoms (weakness) for more than 6 months (inclusive) and less than 36 months(inclusive).
* Slow vital capacity (SVC), measured three times, one of the measure being >/= 70% of that predicted.
* Treated with riluzole at the stable dose of 50 mg bid for at least 30 days before enrolment.

Exclusion Criteria:

* Tracheostomy, invasive ventilation, or non invasive positive pressure ventilation (NIPPV).
* Gastrostomy.
* Evidence of major psychiatric disorder or clinically evident dementia.
* Diagnosis of a neurodegenerative disease in addition to ALS.
* Have a current medication that could interfere with TRO19622 pharmacokinetics: tamoxifene.
* Have current medications that could interfere with TRO19622 absorption such as ezetimibe, bile salts chelators (cholesteramine), fibrates, phytosterols, niacin (vitamin B3),fish oils. Have a current medication of lipid lowering agents other than statins.
* Known hypersensitivity to any component of the study drug.
* Patients with known intolerance or contra-indication to riluzole.
* Have a recent history (within the previous 6 months) or current evidence of alcohol or drug abuse.
* Have concurrent unstable disease involving any system eg, carcinoma other than basal cell carcinoma, any cardiac dysrhythmia, myocardial infarction, clinical or ECG signs of myocardial ischemia, cardiac insufficiency, angina symptoms, current symptoms of Coronary Artery Disease, or any other condition that in the opinion of the Investigator would make the patient unsuitable for study participation.

  . In Germany: Have any cardiac dysrhythmia, myocardial infarction, clinical or ECG signs of myocardial ischemia, cardiac insufficiency, angina symptoms, current symptoms of Coronary Artery Disease or any cardiovascular illness known or identified at the screening or inclusion visits, or have concurrent unstable disease involving any system eg, carcinoma other than basal cell carcinoma or any other condition that in the opinion of the Investigator would make the patient unsuitable for study participation.
* Having a baseline QTc (Bazett) > 450 msec for males and > 470 msec for females.
* Patients with known hepatitis B/C or HIV positive serology.
* Be pregnant female or lactating.
* Have renal impairment defined as blood creatinine > 1:5 X upper limit of normal.
* Have hepatic impairment and/or liver enzymes (ALAT or ASAT) > 3 X ULN.
* Hemostasis disorders or current treatment with oral anticoagulants.
* Be possibly dependent on the Investigator or the Sponsor (eg, including, but not limited to, affiliated employee).
* Participated in any other investigational drug or therapy study with a non approved medication, within the previous 3 months.
* Patients without Social Security Insurance (France).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- University Hospital Gasthuisberg - Dept Neurology - Herestraat 49, Leuven, Belgium
- France (7):
  - HCL Hôpital Neurologique et Neurochirurgical Pierre Wertheimer - Neurologie C et Laboratoire d'électromyographie - 59, boulevard Pinel, Bron
  - CHRU de LILLE - Hôpital Roger Salengro - Centre SLA-MMN - Sce de Neurologie et Pathologie du Mouvement, Lille
  - Centre SLA Limoges - Service de Neurologie, Limoges
  - Hôpital La Timone - Service Neurologie et Maladies Neuromusculaires, Marseille
  - Clinique du Motoneurone - Sce d'Explorations Neurologiques - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nice - Hôpital de l'Archet 1 - Centre de Référence pour les Maladies Neuromusculaires et la SLA, Nice
  - Groupe Hospitalier PITIE-SALPETRIERE - Fédération des Maladies du Système Nerveux, Paris
- Germany (4):
  - Charité Universitätsmedizin Berlin, Campus Virchow-Klinikum, Neurologische Poliklinik Ambulanz für ALS und andere Motoeneuronenerkrankungen, Berlin
  - Universitätsklinik und Poliklinik für Neurologie - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Neurologische Klinik Medizinische Hochschule, Hanover
  - Universitäts- und Rehabilitationskliniken Ulm (RKU) - Neurologische Universitätsklinik, Ulm
- Hospital Carlos III - Unidad de ELA - Sinesio Delgado, 10, Madrid, Spain
- United Kingdom (2):
  - King's MND Care and Research Center - Academic Neurosciences Building PO Box 41 Institute of Psychiatry, London
  - Academic Neurology Unit - University of Sheffield - Section of Neuroscience - Division of Genomic Medicine - School of Medicine and Biomedical Sciences, Sheffield

REFERENCES:
- [Derived] Witzel S, Frauhammer F, Steinacker P, Devos D, Pradat PF, Meininger V, Halbgebauer S, Oeckl P, Schuster J, Anders S, Dorst J, Otto M, Ludolph AC. Neurofilament light and heterogeneity of disease progression in amyotrophic lateral sclerosis: development and validation of a prediction model to improve interventional trials. Transl Neurodegener. 2021 Aug 26;10(1):31. doi: 10.1186/s40035-021-00257-y. PMID 34433481
- [Derived] Devos D, Moreau C, Kyheng M, Garcon G, Rolland AS, Blasco H, Gele P, Timothee Lenglet T, Veyrat-Durebex C, Corcia P, Dutheil M, Bede P, Jeromin A, Oeckl P, Otto M, Meininger V, Danel-Brunaud V, Devedjian JC, Duce JA, Pradat PF. A ferroptosis-based panel of prognostic biomarkers for Amyotrophic Lateral Sclerosis. Sci Rep. 2019 Feb 27;9(1):2918. doi: 10.1038/s41598-019-39739-5. PMID 30814647

RESULTS

PARTICIPANT FLOW:
Groups:
- Olesoxime: 2 capsules of TRO19622 (330mg) once a day with the noon meal as add-on therapy to riluzole 50mg bid.
  Olesoxime: 2 capsules of TRO19622 (330mg) once a day with the noon meal as add-on therapy to riluzole 50mg bid.
  Riluzole: Riluzole given as add-on therapy 50mg bid.
- Placebo Comparator: 2 capsules of Placebo once a day with the noon meal as add-on therapy to riluzole 50mg bid Placebo Comparator: 2 capsules of Placebo once a day with the noon meal as add-on therapy to riluzole 50mg bid Riluzole: Riluzole given as add-on therapy 50mg bid
Period: Overall Study
Arm/Group | Olesoxime | Placebo Comparator
Started | 259 | 253
Completed | 147 | 139
Not Completed | 112 | 114
Not completed — Death | 58 | 65
Not completed — Withdrawal by Subject | 33 | 25
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 9 | 10
Not completed — Lack of efficacy, logistics, unwell | 9 | 10
Not completed — Non-compliance with IMP | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants irrespective of study medication administration and eligibility status.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olesoxime | Placebo Comparator | Total
Number analyzed (Participants) | 259 | 253 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.2) | 55.7 (11.2) | 56.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 89 | 181
  Male | 167 | 164 | 331
Region of Enrollment [Count of Participants; unit: Participants]
  France | 113 | 108 | 221
  Spain | 33 | 34 | 67
  Belgium | 13 | 12 | 25
  Germany | 73 | 74 | 147
  United Kingdom | 27 | 25 | 52

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 18 Months
Description: Overall survival was defined from the date of randomization until the date of death (event) or last known alive date (censored). If the death date was after 18 months, the participant was censored at 18 months (548 days). Participants still alive at or after 18 months were censored at 18 months/ 548 days. All data over the 18-month follow-up period after randomization, and participant survival status at the 18-month follow-up visit for participants who withdrew prematurely from the study for reasons other than death were included.
Time Frame: From the date of randomization until the date of death or last follow-up censored at 18 months (548 days)
Population: ITT population included all randomized participants irrespective of study medication administration and eligibility status.
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
percentage of partcipants | 67.5 [61.0 to 73.1] | 69.4 [63.0 to 74.9]
Statistical Analysis 1: Comparison: Olesoxime vs Placebo Comparator; Test type: Superiority; p = 0.71, Stratified Log-Rank Test

2. Secondary Outcome: Percentage of Participants With Failure Over 18 Months
Description: Time to failure was defined as the time from randomization to the time of the first event to consider (Tracheostomy, invasive ventilation [IV] or non invasive ventilation [NIV])
Time Frame: From randomization to the time of the first event to consider at 18 months (548 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
percentage of participants | 67.1 [60.5 to 72.7] | 65.5 [59.1 to 71.2]
Statistical Analysis 1: Comparison: Olesoxime vs Placebo Comparator; Test type: Superiority; p = 0.83, Stratified Log-Rank Test
Statistical Analysis 2: Comparison: Olesoxime vs Placebo Comparator; Test type: Superiority; p = 0.73, Non-stratified Log-Rank Test

3. Secondary Outcome: Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R)
Description: The ALSFRS-R is an ordinal rating scale (0 through 4) used to determine the ALS participant's self assessment of their ability and need for assistance in 12 activities or functions. This is a validated scale, both in person and by phone, which provides a total score from four sub-scores which assess speech and swallowing, (bulbar function), use of upper extremities (cervical function), gait and turning in bed (lumbar function), and breathing (respiratory function). Total scores range from 0 (most impaired) to 48 (normal ability).
Time Frame: Inclusion, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12, Month 15 and Month 18
Population: ITT population included all randomized participants irrespective of study medication administration and eligibility status. Number analyzed indicates number of participants who were evaluated for the specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
score on a scale
  Inclusion: number analyzed (Participants) | 258 | 251
  Inclusion | 39.1 (4.78) | 38.2 (5.25)
  Month 1: number analyzed (Participants) | 258 | 252
  Month 1 | 38.2 (5.46) | 37.2 (5.59)
  Month 2: number analyzed (Participants) | 247 | 247
  Month 2 | 37.6 (5.64) | 36.7 (6.02)
  Month 3: number analyzed (Participants) | 251 | 242
  Month 3 | 36.4 (6.29) | 35.3 (6.62)
  Month 6: number analyzed (Participants) | 230 | 225
  Month 6 | 34.3 (7.11) | 33.1 (7.62)
  Month 9: number analyzed (Participants) | 205 | 201
  Month 9 | 32.7 (7.72) | 30.4 (8.23)
  Month 12: number analyzed (Participants) | 182 | 175
  Month 12 | 30.5 (8.34) | 28.8 (8.47)
  Month 15: number analyzed (Participants) | 163 | 147
  Month 15 | 28.6 (8.56) | 27.6 (8.92)
  Month 18: number analyzed (Participants) | 148 | 136
  Month 18 | 27.0 (9.38) | 26.3 (9.13)

4. Secondary Outcome: Percentage of Participants With a Global ALS FRS-R Score of <30 or Death
Description: Percentage of participants with a global ALS FRS-R score of < 30 or death was estimated using the Kaplan-Meier method in the ITT, with a two-tailed log-rank, both stratified by site of onset (bulbar or spinal) and non-stratified. The ALSFRS-R is an ordinal rating scale (0 through 4) used to determine the ALS participant's self assessment of their ability and need for assistance in 12 activities or functions. This is a validated scale, both in person and by phone, which provides a total score from four sub-scores which assess speech and swallowing, (bulbar function), use of upper extremities (cervical function), gait and turning in bed (lumbar function), and breathing (respiratory function). Total scores range from 0 (most impaired) to 48 (normal ability).
Time Frame: Month 18 (548 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
percentage of participants | 28.2 [22.5 to 34.1] | 24.9 [19.2 to 30.8]
Statistical Analysis 1: Comparison: Olesoxime vs Placebo Comparator; Test type: Superiority; p = 0.21, Stratified Log-Rank Test
Statistical Analysis 2: Comparison: Olesoxime vs Placebo Comparator; Test type: Superiority; p = 0.20, Non-stratified Log-Rank Test

5. Secondary Outcome: Slow Vital Capacity (SVC) Percent Predicted
Description: SVC as a percent of the predicted value was evaluated and reported.
Time Frame: Baseline, Inclusion, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15 and Month 18
Population: ITT population included all randomized participants irrespective of study medication administration and eligibility status. Number analyzed indicates number of participants who were evaluated at specified time points.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
percentage (%)
  Baseline | 93.1 (14.6) | 93.1 (15.4)
  Month 1: number analyzed (Participants) | 257 | 251
  Month 1 | 89.7 (17.8) | 89.7 (17.6)
  Month 3: number analyzed (Participants) | 249 | 238
  Month 3 | 84.8 (20.4) | 85.7 (19.7)
  Month 6: number analyzed (Participants) | 226 | 219
  Month 6 | 80.7 (22.9) | 80.5 (22.5)
  Month 9: number analyzed (Participants) | 195 | 190
  Month 9 | 77.9 (24.3) | 75.5 (24.7)
  Month 12: number analyzed (Participants) | 170 | 160
  Month 12 | 74.5 (25.4) | 71.3 (29.0)
  Month 15: number analyzed (Participants) | 150 | 150
  Month 15 | 70.5 (28.8) | 71.4 (27.1)
  Month 18: number analyzed (Participants) | 131 | 118
  Month 18 | 69.0 (27.6) | 67.1 (25.5)

6. Secondary Outcome: Percentage of Participants With SVC Percent Predicted <70% or Had Died Over 18 Months
Time Frame: Month 18 (548 days)
Population: ITT population included all randomized participants irrespective of study medication administration and eligibility status. Number analyzed indicates number of participants who were evaluated for specified analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
percentage of participants | 28.9 [23.0 to 35.1] | 31.9 [25.6 to 38.4]
Statistical Analysis 1: Comparison: Olesoxime vs Placebo Comparator; Test type: Superiority; p = 0.56, Stratified Log-Rank Test

7. Secondary Outcome: Global Score of Manual Muscle Testing (MMT) of 34 Muscle Groups
Description: MMT score involved the examination of 30 items. These 30 items are scored from 0 (no trace of contraction) to 5 (normal power at first try). The global score is the sum of the item scores and can range from 0 to 150. Higher score indicates some power.
Time Frame: Inclusion, Month 3, Month 6, Month 9, Month 12, Month 15 and Month 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
score on a scale
  Inclusion: number analyzed (Participants) | 257 | 250
  Inclusion | 128 (18.0) | 126 (18.8)
  Month 3: number analyzed (Participants) | 249 | 239
  Month 3 | 121 (22.8) | 120 (22.0)
  Month 6: number analyzed (Participants) | 226 | 221
  Month 6 | 117 (24.4) | 114 (24.6)
  Month 9: number analyzed (Participants) | 200 | 196
  Month 9 | 112 (27.1) | 109 (27.1)
  Month 12: number analyzed (Participants) | 177 | 168
  Month 12 | 106 (29.7) | 103 (29.6)
  Month 15: number analyzed (Participants) | 159 | 137
  Month 15 | 101 (32.0) | 99.2 (31.2)
  Month 18: number analyzed (Participants) | 147 | 132
  Month 18 | 95.2 (33.7) | 91.8 (34.7)

8. Secondary Outcome: The Single-Item Mc Gill Quality of Life Scale
Description: The single-item McGill quality of life scale evaluated the following question "Considering all parts of my life - physical, emotional, social, spiritual, and financial - over the past two (2) days, the quality of my life has been…"as a score of 1 to 10 on a visual analog scale where 0 is very bad and 10 is excellent.
Time Frame: Inclusion, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15 and Month 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olesoxime | Placebo Comparator
Number analyzed (Participants) | 259 | 253
score on a scale
  Inclusion: number analyzed (Participants) | 257 | 249
  Inclusion | 6.51 (1.65) | 6.47 (1.65)
  Month 1: number analyzed (Participants) | 250 | 245
  Month 1 | 6.17 (1.73) | 6.27 (1.78)
  Month 3: number analyzed (Participants) | 251 | 240
  Month 3 | 5.83 (1.98) | 5.75 (1.89)
  Month 6: number analyzed (Participants) | 229 | 223
  Month 6 | 5.55 (2.12) | 5.50 (2.00)
  Month 9: number analyzed (Participants) | 202 | 197
  Month 9 | 5.30 (2.14) | 5.25 (2.00)
  Month 12: number analyzed (Participants) | 180 | 172
  Month 12 | 4.97 (2.11) | 5.10 (2.02)
  Month 15: number analyzed (Participants) | 161 | 145
  Month 15 | 4.96 (2.26) | 4.90 (2.13)
  Month 18: number analyzed (Participants) | 146 | 132
  Month 18 | 4.77 (2.29) | 5.01 (2.16)

ADVERSE EVENTS:
Time Frame: Safety was assessed during the 18-months study duration.
Description: Clinical and biological safety of TRO19622 co-administered with riluzole were assessed at each visit.
Arm/Group | Olesoxime | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 79/259 | 80/253
Serious Adverse Events (participants affected / at risk) | 68/259 | 65/253
Other Adverse Events (participants affected / at risk) | 98/259 | 101/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olesoxime (N=259) | Placebo Comparator (N=253)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5
Lobar pneumonia (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Device breakage (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 2
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2
Aortic dissection (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1
Areflexia (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Hypercapnic encephalopathy (Nervous system disorders) | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Application site inflammation (General disorders) | 1 | 0
Application site pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2
Renal colic (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Mechanical ventilation (Surgical and medical procedures) | 2 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olesoxime (N=259) | Placebo Comparator (N=253)
Diarrhoea (Gastrointestinal disorders) | 27 | 15
Nausea (Gastrointestinal disorders) | 15 | 16
Bronchitis (Infections and infestations) | 10 | 15
Nasopharyngitis (Infections and infestations) | 22 | 36
Fall (Injury, poisoning and procedural complications) | 26 | 19
Headache (Nervous system disorders) | 19 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 15
Hypertension (Vascular disorders) | 7 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less